CLINICAL TRIAL: NCT03933267
Title: Effects of Cervical Sensorimotor Control Training in Nonspecific Chronic Neck Pain
Brief Title: Cervical Sensorimotor Control Training in Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RiphahIU Aruba Iram
Record Dates: First submitted 2019-04-27; First posted 2019-05-01 (Actual); Last update posted 2019-08-09 (Actual); Status verified 2019-08

CONDITIONS: Nonspecific Chronic Neck Pain
Keywords: Cervical Pain; Kinesthesis
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Intervention Model Description: Both experimental and control groups will be treated simultaneously with one treatment option common to both groups
Who Masked: Participant
Masking Description: This study will be single blinded randomized control trail, participants will be unaware of treatment groups, they will be randomly allocated through sealed envelope method.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Experimental): This group of participant will receive Cervical sensorimotor control training exercises. In addition to it conventional physical therapy protocol will be given.
  Interventions: Other: Cervical sensorimotor control training exercises
- Group II Control (Active Comparator): this group of participant will receive Conventional physical therapy protocol.
  Interventions: Other: Conventional Exercises

INTERVENTIONS:
Other: Cervical sensorimotor control training exercises — Cervical sensory motor training exercises consisting of cervical position sense and cervical movement sense exercises with 3 levels of difficulty and 5 repetitions * 3 sets for each exercise will be given. Some exercises are:
  Head relocation with laser feedback:
  head relocation to neutral and predetermined position with eyes opened (in horizontal / vertical direction) (5 reps x 3 sets) Head relocation to neutral, predetermined and to specific targets with eyes opened (in diagonal directions) (5 reps x 3 sets) Head relocation to neutral and predetermined position with eyes closed (in all directions)(5 reps x 3 sets) In addition to it conventional physical therapy protocol consisting of Generalized stretching and cervical strengthening exercises along with joint mobility.
  Other Names: Prioprioception Exercises
  Arms: Group I
Other: Conventional Exercises — conventional physical therapy protocol consisting of Generalized stretching and cervical strengthening exercises along with joint mobility exercises will be given to patients.
  Arms: Group II Control

SUMMARY:
Impaired cervical joint position sense is associated with neck pain. This study will determine the effects of sensorimotor control training exercises on cervical joint position, pain, ROM and function in nonspecific chronic neck pain. There will be two groups ; experimental and control. Half of study group will receive cervical sensorimotor control training exercises and half of study group will receive conventional physiotherapy protocol.

DETAILED DESCRIPTION:
The study is Randomized Control Trail , which is being conducted in physical therapy Out patient department of Pakistan Railway hospital (April 2019-July 2019) . Sample size of 18 individual was calculated using Epitool with 95% confidence interval (CI), and power 80%. Individual will be screened out according to inclusion criteria. Individuals will be allocated randomly into two groups , 9 in cervical Sensori-motor training group and 9 in conventional physiotherapy protocol group by sealed envelope method.

Both groups will receive conventional physiotherapy protocol (hot pack, stretching exercises and strengthening exercises) for neck pain in common and the experimental group will receive cervical sensorimotor control training in addition to conventional protocol.

Assessment will be done on baseline and 6th week.

Data will be analysed on SPSS version 21.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 to 50 years
* Non specific neck pain
* Insidious neck pain for at least 3 month
* Average pain intensity over the past week >4 on Numeric Pain Rating Scale(NPRS)

Exclusion Criteria:

* Previous history of neck and head trauma or surgery
* Inflammatory joint disease
* Systemic conditions
* Cognitive impairment
* Taking four or more medications

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2019-04-25 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Cervical Joint position error | Baseline
  The task is to return head to the starting position as accurately as possible. Three trials will be performed of right and left rotation and extension. An average absolute error of > 4.5° in any direction is indicative of a deficit in cervical joint position sense
Cervical Joint position error | post 6th week
  The task is to return head to the starting position as accurately as possible. Three trials will be performed of right and left rotation and extension. An average absolute error of > 4.5° in any direction is indicative of a deficit in cervical joint position sense
Clinical test of sensory interaction and balance (CTSIB) | Baseline
  This test is design to assess how well an older adult is using sensory inputs when one or more sensory systems are compromise. Begin timing each trial using a stopwatch. The trial is over when (a) the participant opens his/her eyes in an eyes closed condition, (b) raises arms from sides, (c) loses balance and requires manual assistance to prevent a fall
Clinical test of sensory interaction and balance (CTSIB) | post 6th week
  This test is design to assess how well an older adult is using sensory inputs when one or more sensory systems are compromise. Begin timing each trial using a stopwatch. The trial is over when (a) the participant opens his/her eyes in an eyes closed condition, (b) raises arms from sides, (c) loses balance and requires manual assistance to prevent a fall

SECONDARY OUTCOMES:
Numeric pain rating scale (NPRS) | Baseline
  Numeric pain rating scale (NPRS) is an 11 point (0-10) Scale used to measure pain. Patient verbally select value between (0-10) on the basis of intensity of pain. (0) means No pain and (10) means maximum pain experienced at baseline.
Numeric pain rating scale (NPRS) | post 6th week
  Numeric pain rating scale (NPRS) is an 11 point (0-10) Scale used to measure pain. Patient verbally select value between (0-10) on the basis of intensity of pain. (0) means No pain and (10) means maximum pain experienced at 6th week of intervention.
Neck Disability Index (NDI): | Baseline
  Neck Disability Index (NDI) is a questionnaire designed to assess how neck pain has affected patient's ability to manage in everyday life. It has total 10 sections, For each section the total possible score is 5: if the first statement is marked the section score = 0, if the last statement is marked it = 5. If all ten sections are completed the score is calculated and converted into percentages. The maximum Score of Neck Disability Index (NDI) is 50. It is measured at Baseline before Intervention.
Neck pain and disability index (NDI): | post 6th week
  Neck Disability Index (NDI) is a questionnaire designed to assess how neck pain has affected patient's ability to manage in everyday life. It has total 10 sections, For each section the total possible score is 5: if the first statement is marked the section score = 0, if the last statement is marked it = 5. If all ten sections are completed the score is calculated and converted into percentages. The maximum Score of Neck Disability Index (NDI) is 50. It is measured after 6th week of Intervention.
CROM (inclinometer) | Baseline
  A cervical range of motion (CROM) inclinometer will be use to assess cervical range of motion in flexion, extension, left right lateral flexion and left-right rotation. Participants will be seated upright and asked to actively move their neck in each direction.
CROM (inclinometer) | post 6th week
  A cervical range of motion (CROM) inclinometer will be use to assess cervical range of motion in flexion, extension, left right lateral flexion and left-right rotation. Participants will be seated upright and asked to actively move their neck in each direction.
Patient-Specific Functional Scale (PSFS) | baseline
  The patient-specific functional scale (PSFS) will be use to assess participants' functional status. Participants will be ask to nominate 3 to 5 activities that they are unable to do or having difficulty doing because of their neck pain. These activities will be rated on a 0-10 scale, where 0 is unable to perform the activity and 10 is able to perform the activity at same. An average of all activities scores will be use for analysis
Patient-Specific Functional Scale (PSFS) | post 6th week
  The patient-specific functional scale (PSFS) will be use to assess participants' functional status. Participants will be ask to nominate 3 to 5 activities that they are unable to do or having difficulty doing because of their neck pain. These activities will be rated on a 0-10 scale, where 0 is unable to perform the activity and 10 is able to perform the activity at same. An average of all activities scores will be use for analysis

CONTACTS AND LOCATIONS:
Overall Officials: Huma Riaz, PHD*, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Railway hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Javanshir K, Ortega-Santiago R, Mohseni-Bandpei MA, Miangolarra-Page JC, Fernandez-de-Las-Penas C. Exploration of somatosensory impairments in subjects with mechanical idiopathic neck pain: a preliminary study. J Manipulative Physiol Ther. 2010 Sep;33(7):493-9. doi: 10.1016/j.jmpt.2010.08.022. PMID 20937427
- [Background] Saadat M, Salehi R, Negahban H, Shaterzadeh MJ, Mehravar M, Hessam M. Postural stability in patients with non-specific chronic neck pain: A comparative study with healthy people. Med J Islam Repub Iran. 2018 Apr 23;32:33. doi: 10.14196/mjiri.32.33. eCollection 2018. PMID 30159284
- [Background] de Vries J, Ischebeck BK, Voogt LP, van der Geest JN, Janssen M, Frens MA, Kleinrensink GJ. Joint position sense error in people with neck pain: A systematic review. Man Ther. 2015 Dec;20(6):736-44. doi: 10.1016/j.math.2015.04.015. Epub 2015 May 2. PMID 25983238
- [Background] Beinert K, Taube W. The effect of balance training on cervical sensorimotor function and neck pain. J Mot Behav. 2013;45(3):271-8. doi: 10.1080/00222895.2013.785928. PMID 23663191
- [Background] Swait G, Rushton AB, Miall RC, Newell D. Evaluation of cervical proprioceptive function: optimizing protocols and comparison between tests in normal subjects. Spine (Phila Pa 1976). 2007 Nov 15;32(24):E692-701. doi: 10.1097/BRS.0b013e31815a5a1b. PMID 18007229